CLINICAL TRIAL: NCT02700061
Title: Effects of Upper Limb Motor Training and Upper Limb Robotic Training Over Neuroplasticity and Function Capacity: A Single-blind Randomized Clinical Trial With Patients With Stroke Sequelae
Brief Title: Effects of Upper Limb Motor and Robotic Training Over Neuroplasticity and Function Capacity
Acronym: NARLE1
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 0910.0.015.000-11
Record Dates: First submitted 2015-11-24; First posted 2016-03-07 (Estimated); Last update posted 2016-03-07 (Estimated); Status verified 2015-08

CONDITIONS: Stroke
Keywords: Induced Constraint Therapy; Robotic Occupational Therapy; Neuroplasticity
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Induced Constraint Therapy - ICT (Experimental): Physical rehabilitation with Induced Constraint Therapy as part of the occupational therapy. Standard Occupational Therapy two times a week for ten weeks, followed by two whole weeks of Induced Constraint Therapy.
  Interventions: Procedure: Induced Constraint Therapy - ICT
- Robotic occupational therapy (Experimental): Physical rehabilitation with Robotic occupational therapy. Robotic Occupational Therapy three times a week for twelve weeks.
  Interventions: Procedure: Robotic occupational therapy

INTERVENTIONS:
Procedure: Robotic occupational therapy — Robotic Occupational Therapy three times a week for twelve weeks.
  Other Names: Robotic therapy
  Arms: Robotic occupational therapy
Procedure: Induced Constraint Therapy - ICT — Standard Occupational Therapy two times a week for ten weeks, followed by two whole weeks of Induced Constraint Therapy.
  Other Names: ICT
  Arms: Induced Constraint Therapy - ICT

SUMMARY:
The purpose of this study is to evaluate and compare the effects of upper limb training with Induced Constraint Therapy (ICT) or robotic therapy. No placebo therapy is used. Motor function, neurological evaluations and quality of life are assessed for the comparison of the therapies.

DETAILED DESCRIPTION:
The trial is being carried out in the Institute of Physical Medicine and Rehabilitation of the University of São Paulo since February 2012. The investigators are including patients with clinical diagnosis of Ischemic or hemorrhagic stroke.

The patients are being randomized in blocks of four, six and eight, in two arms: ICT: patients are undergoing 60 minutes physiotherapy and occupational therapy twice a week for ten consecutive weeks. Other therapeutic services as phonoaudiology, psychology, nutrition, physical conditioning are prescribed upon the patients' medical demands. After the 10 weeks, the patients are undergoing two whole weeks of daily ICT as to reach 90% of the time under constraint, including weekends. During this last period, no other therapeutic service is offered, but the occupational therapy under ICT. Patients are not allowed to undergo robotic therapy.

Robotic therapy: patients are undergoing robotic occupational therapy for 60 minutes, three times a week for twelve consecutive weeks. All other therapeutic services are prescribed upon the patients' medical demands. Patients are not allowed to undergo ICT.

The investigator and the raters are blind to treatment.

The evaluations are done prior to the beginning of the treatment and at the end of it. The follow up assessments are done at 3 and 12 months after the end of the treatment.

The sample size was estimated to be 62 patients in each arm, a total size of 124 patients

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of stroke;
* Patients from 6 months after stroke up to 36 months after stroke;
* Clinically stable;
* Upper limb Brunnstrom scale III or IV;
* Brunnstrom scale above V if clinician supports patients will benefit from treatment;
* Minimum wrist extension of 20°, and minimum of 10° of metacarpophalangeal active extension.
* Signed Informed Consent Form;

Exclusion Criteria:

* Mini-Mental score lower than 20 points;
* Previous multiple strokes;
* Bone diseases and articulation injuries ;
* Presence of psychological disturbances capable of diminishing adherence;
* Articulation pain within the range of motion proposed by the therapies;
* Participation in another study protocol for upper limbs therapies.
* Previous treatment with robotic assisted therapies.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2012-02; Primary Completion 2016-04 (Estimated); Study Completion 2017-02 (Estimated)

PRIMARY OUTCOMES:
Change on Motor Function assessed by Wolf Motor Function scale | Baseline and 12 weeks
  Change from baseline in Wolf Motor Function scale.
Change on Motor Function assessed by Fugl Meyer scale | Baseline and 12 weeks
  Change from baseline in Fugl Meyer scale.

SECONDARY OUTCOMES:
Change on Motor Function assessed by Wolf Motor Function scale | Baseline, 3 months and 12 months
  Multiple changes from baseline in Wolf Motor Function scale.
Change on Motor Function assessed by Fugl Meyer scale | Baseline, 3 months and 12 months
  Multiple changes from baseline in Fugl Meyer scale.
Change on Motor Function assessed by Robotic scale | Baseline, 3 months and 12 months
  Multiple changes from baseline in robotic scale.
Change on Function ability and quality of movement assessed by Arm Motor Ability Test (AMAT) | Baseline, 12 weeks, 3 months and 12 months
  Multiple changes from baseline in AMAT scale.
Change on Functional Independence Measure (FIM) as assessed by FIM scale | Baseline, 12 weeks, 3 months and 12 months
  Multiple changes from baseline in FIM scale.
Change on Quality of life assessed by Stroke Impact Scale (SIS) | Baseline, 12 weeks, 3 months and 12 months
  Multiple changes from baseline in SIS.
Change on Kinematic variables assessed by InMotion robots | Baseline, 12 weeks, 3 months and 12 months
  Multiple motion changes from baseline in the Kinematic variables assessed by InMotion robots.

OTHER OUTCOMES:
Psychological Evaluation assessed by Perceived Stress Scale (PSS-10) | Baseline, 12 weeks, 3 months and 12 months
  Multiple changes from baseline in PSS-10.
Neuroplasticity as assessed by Brain Derived Neurotrophic Factor (BDNF) | Baseline, 12 weeks, 3 months and 12 months
  Multiple changes from baseline in BDNF.
Corticospinal excitability as assessed by transcranial magnetic stimulation (TMS) | Baseline, 12 weeks, 3 months and 12 months
  Multiple changes from baseline in TMS.
Neurologic evaluation as assessed by electroencephalography | Baseline, 12 weeks, 3 months and 12 months
  Multiple changes from baseline in electroencephalography.

CONTACTS AND LOCATIONS:
Overall Officials: Linamara Rizzo Battistella, Md PhD, Principal Investigator — University of Sao Paulo
Locations (1):
- Centro de Pesquisa Clínica do Instituto de Medicina Física e Reabilitação do HCFMUSP, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Terranova TT, Simis M, Santos ACA, Alfieri FM, Imamura M, Fregni F, Battistella LR. Robot-Assisted Therapy and Constraint-Induced Movement Therapy for Motor Recovery in Stroke: Results From a Randomized Clinical Trial. Front Neurorobot. 2021 Jul 21;15:684019. doi: 10.3389/fnbot.2021.684019. eCollection 2021. PMID 34366819